CLINICAL TRIAL: NCT06301425
Title: Measurable Residual Disease Response-adapted Allogeneic Hematopoietic Stem Cell Transplantation for Adverse-risk Acute Myeloid Leukemia: an Open-label, Randomized, Controlled Trial（TROPHY-AML01）
Brief Title: MRD Response-adapted Allo-HSCT for Adverse-risk AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Ruijin Hospital (Other); Wuhan TongJi Hospital (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Director, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROPHY-AML01
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Allogeneic hematopoietic stem cell transplantation; Measurable residual disease; Adverse risk
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): According to the MFC MRD status after the first consolidation (MRDcon1), the MRDcon1 positive patients were categorized into high-risk group (i.e., risk stratification). All the patients in high-risk group who fulfilled all inclusion/exclusion criteria were randomly assigned in a 1:1 ratio to receive a second consolidation therapy (intervention group) or receive allo-HSCT directly (control group).
  Interventions: Other: Intervention group
- Control group (Active Comparator): According to the MFC MRD status after the first consolidation (MRDcon1), the MRDcon1 positive patients were categorized into high-risk group (i.e., risk stratification). All the patients in high-risk group who fulfilled all inclusion/exclusion criteria were randomly assigned in a 1:1 ratio to receive a second consolidation therapy (intervention group) or receive allo-HSCT directly (control group).
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention group — Patients in interventional group could choose one of the following treatment protocols and then receive allo-HSCT if they were CR after the second consolidation:
  1. . Venetoclax plus azacitidine: azacitidine 75mg/m2/d d1-7; venetoclax 400mg/d, d1-21;
  2. . Venetoclax plus CAG: venetoclax 400mg qd d1-14; aclacinomycin 20mg qd d1-4; cytarabine 10mg/m2 q12h subcutaneous injection d1-14; G-CSF 300μg qd d1-14;
  3. . Venetoclax plus IA: venetoclax 400mg qd d1-4; idarubicin 10mg qd d1-4; cytarabine 500mg qd d1-4;
  4. . Venetoclax plus AA: venetoclax 400mg qd d1-7; aclacinomycin 20mg qd d1-7; cytarabine 100mg/m2 qd d1-7.
  Arms: Intervention group
Other: Control group — Receive allo-HSCT directly without the second consolidation chemotherapy.
  Arms: Control group

SUMMARY:
This TROPHY-AML01 regimen aims to identify the effectiveness and safety of MRD response-adapted allo-HSCT for adverse-risk acute myeloid leukemia in an open-label, randomized, controlled trial.

DETAILED DESCRIPTION:
1.1 Relapse is the most important cause of transplant failure Acute myeloid leukemia is one the most important hematologic malignancies for adults. According to the criteria of European LeukemiaNet (ELN) 2022, approximately 40%-50% of AML patients were categorized into adverse-risk group. The clinical outcomes of these patients receiving chemotherapy alone is poor and the 4-year probability of leukemia-free survival (LFS) after therapy is nearly 10%. Thus, allogeneic hematologic stem cell transplantation (allo-HSCT) is considered as the critical consolidation in adverse-risk AML patients, and many AML patients could achieve long-term LFS after allo-HSCT. However, nearly one third of the adverse-risk AML patients would experience relapse after allo-HSCT, and the outcomes of patients with post-transplant are very poor and relapse is also the most important cause of mortality after allo-HSCT. Thus, how to prevent post-transplant relapse is important to further improve the survival of patients with adverse-risk AML.

1.2 Measurable residual disease (MRD) can predict the relapse of AML after treatment.

The detection of MRD is one of the most important methods for defining the depth of remission. Using current sensitive techniques, the presence of 1 residual leukemia cell in 10 000-1 000 000 cells can be detected in patients with morphological complete remission (CR). The most commonly used method for MRD assessment involves (1) the determination of leukemia-associated immunophenotypic patterns (LAIPs) using multiparameter flow cytometry (MFC) and (2) the quantitative polymerase chain reaction (qPCR)-based evaluation of expression levels of leukemia-related genes, such as recurrent genetic abnormalities and other mutation types.

1.3 Pre-transplant MRD can predict the relapse of AML after allo-HSCT. MFC is one of the most common methods for MRD monitoring and is the most important method for MRD monitoring for those without leukemia-specific molecular markers. In the systemic review of Buckley et al., pre-transplant MRD was associated with worse LFS (hazard ratio [HR] = 2.76 [1.90-4.00]), overall survival (OS, HR = 2.36 [1.73-3.22]), and cumulative incidence of relapse (HR = 3.65 [2.53-5.27]).

1.4 The prognostic value of pre-transplant MRD positivity is controversial in adverse-risk AML.

Pre-transplant MRD positivity could predict relapse after allo-HSCT, however, its prognostic value may be more significantly in patients with favorite- and intermediate-risk group. Some authors suggested that pre-transplant MFC MRD was less important in predicting relapse than variables reflecting the biology of the disease (e.g., cytogenetics, molecular marker, or chemotherapy refractory). Receiving repeated consolidation to achieve pre-transplant MRD negativity may not decrease the risk of relapse and improve survival, and patients may experience relapse during consolidation chemotherapy and may suffer additional therapeutic toxicities which may increase the risk of non-relapse mortality after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed AML;
2. Categorized into adverse-risk group according to ELN 2022 criteria;
3. 16-65 years of age at the time of diagnosis;
4. achieving CR after 1 or 2 courses of induction chemotherapies;

4) ECOG PS score of 0 to 1 5) It needs consent from the patients or/and legal guardian, and signature on the Informed Consent.

Exclusion Criteria:

1. Newly diagnosed AML, but categorized into favorite- or intermediate-risk group according to ELN 2022 criteria;
2. < 16 years, or older than 65 years at the time of diagnosis;
3. Achieving CR after 3 or more courses of induction chemotherapies, or could not achieve CR after induction chemotherapies;
4. ECOG PS score of 2 or more;
5. Patients with other comorbidities or mental diseases that influence the life safety and compliance of patients as well as affect informed consent, enrollment in the research, follow-up visit or result interpretation.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 1 year
  EFS, defined as the time from the date of randomization to the date of MRD positivity, relapse, or death due to any cause.

SECONDARY OUTCOMES:
Relapse | 1 year
  Relapse, defined as the time from date of randomization to date of leukemia relapse.
Leukemia-free survival (LFS) | 1 year
  LFS, defined as the time from the date of randomization to the date of relapse or death due to any cause.
Non-relapse mortality (NRM) | 1 year
  NRM, defined as the time from date of randomization to date of death not preceded by leukemia relapse.
Overall survival (OS) | 1 year
  OS, defined as the time from the date of randomization to the date of death due to any cause.
Acute graft-versus-host disease (aGvHD) | 1 year
  aGvHD, defined as the diagnosis of any aGvHD including grade I to IV.
Chronic graft-versus-host disease (cGvHD) | 1 year
  cGvHD, defined as the diagnosis of any cGvHD including mild, moderate, severe.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Mo, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China